CLINICAL TRIAL: NCT03337763
Title: A Multi-center Prospective Pilot Study to tEst LEft Ventricular Intra-cardiac Conduction Time as a Predictor of CRT Response
Brief Title: A Prospective Pilot Study (BIO|SELECT Pilot)
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: CR023
Record Dates: First submitted 2017-10-24; First posted 2017-11-09 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: LV-LV conduction delay
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrolled patients implanted with Biotronik CRT-D and QP lead equipped with MultiPole pacing mode is grouped into which programmed into MultiPole pacing, or conventional bi-ventricular pacing mode. They are followed up by seven month post implantation, and predefined cardiac functional parameters are collected at each visit.

DETAILED DESCRIPTION:
Enrolled patients will undergo the baseline medical tests to assess the cardiac functions (e.g. echo, blood test, and 12-Lead ECG) prior to the implantation of Biotronik CRT-D and QP lead featured with MultiPole Pacing parameter. At implantation, LV-LV conduction delays are measured in predefined LV pacing and sensing configurations. One month after the successful implantation, the patients revisit the investigation site to be adjudicated for programming MultiPole pacing or continuing bi-ventricular pacing mode, based on their echo readings by then. Patients are subsequently followed up at four and seven month post implantation to acquire the LV-LV conduction delays and echo readings, etc. at the time.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study enrollment, candidate patients must meet all of the following criteria

* Indicated for a CRT-D implantation
* Has never received CRT
* Planned to be implanted with a quadripolar LV Lead, and CRT-D with MultiPole pacing feature, both manufactured by BIOTRONIK
* Geographically stable and willing to comply with the required follow-up schedule
* With written informed consent

Exclusion Criteria:

Candidate patients will not be eligible if either of the following criteria is applicable

* Underwent a cardiac surgery within last 3 months, or scheduled for cardiac surgery other than CRT implantation
* Life expectancy is less than a year
* Can not be programmed to MultiPole pacing "ON"
* Does not agree to the concept of HomeMonitoring System
* With known pregnancy
* At age below 20 years
* Participated in another interventional clinical study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with known pregnancy is not eligible
Study Population: The patient collective consists of heart failure patients with CRT-D indication according to clinical routine. Two hundred patients with successful device implantation will be enrolled in the clinical investigation.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Correlation between LV-LV/RV-LV intra-cardiac conduction time and multiple hemodynamic parameters | through study completion, an average of 7 months
  LV-LV/RV-LV intra-cardiac conduction time will be obtained at each time frame, and correlation will be investigated with variation of multiple hemodynamic parameters from baseline up to seven month follow up.

SECONDARY OUTCOMES:
Rate of arrhythmia episodes | through study completion, an average of 7 months
  Comparison between patient groups in terms of rate of arrhythmia
Influence by baseline characteristics | through study completion, an average of 7 months
  An alanysis of the impact of the baseline characteristics on other outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Kyorin University Hospital, Mitaka, Tokyo, Japan